CLINICAL TRIAL: NCT03058666
Title: Comparison of Aerosol Delivery of Infasurf to Usual Care in Spontaneously Breathing RDS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ONY (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aero-02
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: Aerosol; surfactant; calfactant; Infasurf; Respiratory Distress Syndrome; RDS; Premature; Neonates
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — calfactant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Aerosolized Calfactant (Experimental): 1. NICU Patients with a clinical diagnosis of RDS
  2. Inspired oxygen ≥21% to maintain adequate oxygen saturation
  3. Not Intubated
  4. Requiring Nasal continuous positive airway pressure
  Interventions: Drug: Aerosolized Calfactant; Device: Solarys
- Usual Care (No Intervention): There will be no protocol driven interventions in the usual care group.

INTERVENTIONS:
Drug: Aerosolized Calfactant — Aerosolization of Infasurf at 6ml/kg via the modified Solarys aerosol generator.
  Other Names: Infasurf; Calfactant
  Arms: Aerosolized Calfactant
Device: Solarys — Aerosolization of Infasurf at 6ml/kg via the modified Solarys aerosol generator.
  Arms: Aerosolized Calfactant

SUMMARY:
Study to test the hypothesis that aerosolized Infasurf can decrease the need for intubation and instillation of liquid surfactant to the airway.

DETAILED DESCRIPTION:
Treatment will not be masked. The study objective is to document that aerosolized Infasurf is superior to "usual care" and provides for some patients effective surfactant therapy with less need for endotracheal intubation and instillation of a surfactant suspension into the airway. Two cohorts will be recruited: (a) patients who did not receive surfactant at birth who develop RDS in the first hours of life and (b) patients who received instillation of surfactant for RDS in the first hour of life, were extubated, and have continuing RDS.

ELIGIBILITY:
Inclusion Criteria:

RDS Patients

1. NICU patient, ≥1hour of age and <24 hours of age.
2. Clinical diagnosis of RDS, with or without chest X-ray data.
3. Inspired oxygen ≥21% to maintain adequate oxygen saturation.
4. Not intubated
5. Requiring:

   1. nasal continuous positive airway pressure (nCPAP).

Exclusion Criteria:

1. Congenital anomaly limiting care options or requiring early surgery.
2. Cardiopulmonary decompensation.

   1. hypotension with metabolic acidosis (base excess < -10 meq/l).
   2. Oxygen saturations < 88% at start of aerosolization.
   3. PaCO2 ≥ 60 mmHg at start of aerosolization.
3. Grade 3 or Grade 4 intraventricular hemorrhage by cranial ultrasound, if known.
4. Acute hypoxic encephalopathy with or without seizures.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Chair — Albany Medical College
Locations (22):
- United States (22):
  - USA Children's & Women's Hospital, Mobile, Alabama
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Baptist Hospital of Miami, Miami, Florida
  - Adventist Healthcare System, Florida Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - University of South Florida, Tampa general, Tampa, Florida
  - Columbus Regional Hospital, Columbus, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Kentucky Children's Hospital, University of Kentucky Medical Center, Lexington, Kentucky
  - Children's Hospital and Clinics, Minneapolis, Minnesota
  - Children's Hospital Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Sisters of Charity Hospital, Buffalo, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - The Medical University of South Carolina, Charleston, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt university Medical Center, Nashville, Tennessee
  - North central Baptist Hospital, San Antonio, Texas
  - Timpanogos Regional Medical Center, Orem, Utah
  - Utah Valley Hospital, Provo, Utah
  - University of Virgina Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cummings JJ, Gerday E, Minton S, Katheria A, Albert G, Flores-Torres J, Famuyide M, Lampland A, Guthrie S, Kuehn D, Weitkamp JH, Fort P, Abu Jawdeh EG, Ryan RM, Martin GC, Swanson JR, Mulrooney N, Eyal F, Gerstmann D, Kumar P, Wilding GE, Egan EA; AERO-02 STUDY INVESTIGATORS. Aerosolized Calfactant for Newborns With Respiratory Distress: A Randomized Trial. Pediatrics. 2020 Nov;146(5):e20193967. doi: 10.1542/peds.2019-3967. Epub 2020 Oct 15. PMID 33060258

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerosolized Calfactant: 1. NICU Patients with a clinical diagnosis of RDS
  2. Inspired oxygen ≥21% to maintain adequate oxygen saturation
  3. Not Intubated
  4. Requiring Nasal continuous positive airway pressure
  Aerosolized Calfactant: Aerosolization of Infasurf at 6ml/kg via the modified Solarys aerosol generator.
  Solarys: Aerosolization of Infasurf at 6ml/kg via the modified Solarys aerosol generator.
Period: Overall Study
Arm/Group | Aerosolized Calfactant | Usual Care
Started | 241 | 236
Completed | 241 | 236
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 477 were randomized into the two cohorts between April 2017 and June 2018. Having reached our sample size target for cohort 1, further enrollment into cohort 2 was discontinued.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerosolized Calfactant | Usual Care | Total
Number analyzed (Participants) | 241 | 236 | 477
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 241 | 236 | 477
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 33.2 (3.2) | 33.1 (3.1) | 33.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 95 | 195
  Male | 141 | 141 | 282
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 241 | 236 | 477

OUTCOME MEASURES:

1. Primary Outcome: Intubation and Instillation of Liquid Surfactant
Description: Percent of at risk subjects receiving endotracheal intubation and instillation of surfactant within the first 72 hours.
Time Frame: 72 hours
Population: All enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Calfactant | Usual Care
Number analyzed (Participants) | 241 | 236
Participants | 69 | 120

2. Secondary Outcome: Respiratory Support Requirements
Description: Difference of Respiratory support at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Calfactant | Usual Care
Number analyzed (Participants) | 241 | 236
Participants | 65 | 124

3. Secondary Outcome: Air Leak
Description: Percent of at risk subjects with air leak at any time
Time Frame: 28 days
Population: All Enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Aerosolized Calfactant | Usual Care
Number analyzed (Participants) | 241 | 236
Participants | 14 | 11

ADVERSE EVENTS:
Time Frame: Birth to 28 days or discharge, whichever came first.
Arm/Group | Aerosolized Calfactant | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/241 | 1/236
Serious Adverse Events (participants affected / at risk) | 13/241 | 14/236
Other Adverse Events (participants affected / at risk) | 225/241 | 219/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Calfactant (N=241) | Usual Care (N=236)
Air Leak (Respiratory, thoracic and mediastinal disorders) | 13 (23) | 14 (23)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Cardiac disorders) | 6 (6) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spontaneous intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotizing enterocolitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Intraventricular hemorrhage, Grade IV (Nervous system disorders) | 0 (0) | 2 (2)
Periventricular leukomalacia (Nervous system disorders) | 0 (0) | 2 (2)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Primary pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pink colored oral discharge secretion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Calfactant (N=241) | Usual Care (N=236)
Anemia (Blood and lymphatic system disorders) | 53 (53) | 54 (54)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Polycythemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16) | 12 (12)
Bradycardia (Cardiac disorders) | 7 (7) | 6 (6)
Hypotension (Cardiac disorders) | 5 (5) | 4 (4)
Patent ductus arteriosus (Cardiac disorders) | 25 (25) | 27 (27)
Hyperbilirubinemia (Hepatobiliary disorders) | 195 (195) | 191 (191)
Hypocalcemia (Endocrine disorders) | 11 (11) | 13 (13)
Hypophosphatemia (Endocrine disorders) | 5 (5) | 1 (1)
Conjunctivitis (Eye disorders) | 4 (4) | 1 (1)
Retinopathy of prematurity (Eye disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 47 (47) | 37 (37)
Emesis (Gastrointestinal disorders) | 8 (8) | 9 (9)
Feeding Intolerance (Gastrointestinal disorders) | 9 (9) | 9 (9)
Gastroesophageal reflux (Gastrointestinal disorders) | 13 (13) | 9 (9)
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 5 (5) | 2 (2)
Unspecified nutritional deficiency (Gastrointestinal disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 12 (12) | 7 (7)
Sepsis (Infections and infestations) | 14 (14) | 33 (33)
Alkaline phosphatase increase (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (12) | 7 (7)
Hypernatremia (Metabolism and nutrition disorders) | 20 (20) | 16 (16)
Hypochloremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 31 (31) | 38 (38)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 26 (26) | 24 (24)
Metabolic acidosis (Metabolism and nutrition disorders) | 16 (16) | 13 (13)
Apnea (Nervous system disorders) | 116 (116) | 108 (108)
Intraventricular hemorrhage grade I (Nervous system disorders) | 5 (5) | 2 (2)
Intraventricular hemorrhage grade II (Nervous system disorders) | 10 (10) | 3 (3)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 17 (17)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary interstitial emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 14 (14)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Diaper Rash (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Hypovolemia (Vascular disorders) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03058666/Prot_SAP_000.pdf